CLINICAL TRIAL: NCT00349882
Title: Effects of Contact Lens Care Regimens on the Corneal Epithelium
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Waterloo (Other)
Collaborators: Alcon Research (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: P/216/05/L
Record Dates: First submitted 2006-07-05; First posted 2006-07-10 (Estimated); Last update posted 2006-07-10 (Estimated); Status verified 2006-07

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia | interventions — Contact Lenses, Hydrophilic

INTERVENTIONS:
Device: soft contact lens
Drug: Marketed multipurpose disinfection regimen

SUMMARY:
The purpose of this study is to compare the performance of two different contact lens care solutions, specifically their affects on the front surface of the eye.

ELIGIBILITY:
Inclusion Criteria:

1. Is at least 18 years old and has full legal capacity to volunteer.
2. Has read, understood and signed an Information Consent Letter.
3. Is willing and able to follow instructions and maintain the appointment schedule.
4. Is correctable to a visual acuity of 6/6 or better (each eye), with their habitual visual correction.
5. Has normal binocular vision (no strabismus, no amblyopia, and anisometropia less than or equal to 1.00 D).
6. Has clear corneas and no active ocular disease.
7. Has had an ocular examination in the last 2 years.
8. Has not worn contact lenses before, or has worn contact lenses only for a trial period, with no trials occurring within the last six months.

   An ineligible contact lens wearer is one who:
9. Responds positively to points 1 to 7 above.
10. Has a distance contact lens prescription between -0.50D and -9.00 D.
11. Has astigmatism less than or equal to -1.00D cyl.
12. Currently wears silicone hydrogel contact lenses successfully.
13. Agrees to wear the study lenses on a daily wear basis without the use of ocular or lens lubricants.

Exclusion Criteria:

1. Has undergone corneal refractive surgery.
2. Is aphakic.
3. Has any active ocular disease.
4. Has any systemic disease affecting ocular health.
5. Is using any systemic or topical medications that may affect ocular health.
6. Has known sensitivity to the diagnostic pharmaceuticals to be used in the study.
7. Is pregnant or lactating.
8. Is participating in any other type of clinical or research study.

   An ineligible contact lens wearer is one who:
9. Responds positively to any of points 1 to 8 above for exclusion criteria.
10. Has known sensitivity to the contact lens care solutions used in the study.
11. Has ocular or systemic allergies that could adversely affect contact lens wear.
12. Has any ocular pathology or severe insufficiency of lacrimal secretion (dry eyes) that would affect the wearing of contact lenses.
13. Has pinguecula/pterygium that in the investigator's judgement makes contact lens wear inadvisable.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2005-06

PRIMARY OUTCOMES:
The primary outcome measure of this study is to investigate the effects of two
different contact lens care solutions on the cornea.

SECONDARY OUTCOMES:
The secondary outcome measure of this study is to compare the subjective and
objective responses between two different contact lens care solutions.

CONTACTS AND LOCATIONS:
Overall Officials: Craig Woods, PhD, Principal Investigator — University of Waterloo; Desmond Fonn, MOptom, Principal Investigator — University of Waterloo
Locations (1):
- Centre for Contact Lens Research, University of Waterloo, Waterloo, Ontario, Canada